CLINICAL TRIAL: NCT02215811
Title: Treatment of Severe Acute Respiratory Distress Syndrome With Allogeneic Bone Marrow-derived Mesenchymal Stromal Cells
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Karl-Henrik Grinnemo, MD, PhD, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC-ARDS
Record Dates: First submitted 2014-04-11; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Acute Respiratory Distress Syndrome, Adult
Keywords: Extracorporeal membrane oxygenation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mesenchymal stromal cells (Experimental)
  Interventions: Biological: Mesenchymal stromal cells

INTERVENTIONS:
Biological: Mesenchymal stromal cells

SUMMARY:
This is a multi-center, open-label, non-randomized controlled trial. Patients with viral-induced acute respiratory distress syndrome (ARDS) on extracorporeal membrane oxygenation (ECMO) will be eligible. Ten patients will be enrolled and receive allogeneic bone marrow-derived mesenchymal stromal cells (BM-MSC). Ventilator parameters as well as preoperative clinical characteristics and postoperative clinical outcomes will be registered. Routine blood sampling, radiography, and bronchioalveolar lavage will be performed pre- and postoperatively. Spirometry, quality of life assessment, and 6 minute walk test will be performed postoperatively. All available data will be collected prospectively. Follow-up is 12 months. Informed consent will be obtained from relatives to patients meeting the inclusion criteria before the initiation of any study-specific procedures.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Viral-induced acute respiratory distress syndrome
* Ventilator treatment
* Extracorporeal membrane oxygenation treatment
* Relatives provide written informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | During hospital stay, an expected average 2 months

SECONDARY OUTCOMES:
Pulmonary compliance | During ventilator treatment, an expected average of 1 month
Pulmonary tidal volume | During ventilator treatment, an expected average of 1 month
Adverse events | 6 months
  I.e infection, fever, effect on end-organ function
All-cause mortality | 12 months
Recovery of organ functions | 12 months
  kidney, liver, heart functions

OTHER OUTCOMES:
Immune modulation | 3 months
  Change in T-cell, mononuclear cell, cytokine ans microRNA response towards an immunomodulatory phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Henrik Grinnemo, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala